CLINICAL TRIAL: NCT04268134
Title: Omega-3 Fatty Acids, Oxylipins, and Tolerance of Aromatase Inhibitor Therapy
Brief Title: Altering Lipids for Tolerance of Aromatase Inhibitor Therapy
Acronym: ALTA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2019.125; HUM00171150 (Other: University of Michigan)
Record Dates: First submitted 2020-01-29; First posted 2020-02-13 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: Aromatase inhibitor; Omega-3 fatty acid
MeSH Terms: conditions — Breast Neoplasms | interventions — Omacor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Omega 3 fatty acid supplement (Experimental): Omega-3 ethyl esters orally daily (containing 465 mg eicosapentaenoic acid [EPA] and 375 mg docosahexaenoic acid [DHA] per capsule,supplied as 4 x 1gm capsule)
  Interventions: Dietary Supplement: Omega-3 fatty acid supplement

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acid supplement — 4 capsules taken by mouth each day for 24 weeks (starting at the week 12 visit).
  Other Names: Lovaza

SUMMARY:
Aromatase inhibitor medications have been approved by the U.S Food and Drug Administration (FDA) for treatment of hormone receptor positive breast cancer. This treatment has been shown to be very effective for treating breast cancer. However, some patients have difficulty tolerating the treatment, and some even decide to stop treatment because of the side effects. Research has shown that over half of patients who had joint pain and stiffness when taking an aromatase inhibitor had an improvement in their symptoms when they took omega-3 fatty acid supplements. This study is being conducted to test whether having patients start to take an omega-3 fatty acid supplement soon after they starting taking an aromatase inhibitor medicine will reduce the likelihood that they will have bothersome symptoms.

ELIGIBILITY:
Inclusion Criteria

* Female subject aged ≥ 18 years who are postmenopausal according to standard clinical criteria or who will have been receiving LHRH agonist therapy for at least 28 days prior to AI initiation.
* Stage 0-3 estrogen receptor positive (≥1%) and/or progesterone receptor positive (≥1%) breast cancer, or patients at high risk of developing breast cancer who are planning to initiate AI therapy for chemoprevention.
* Planned initiation of aromatase inhibitor therapy (anastrozole, exemestane, or letrozole) for adjuvant treatment of breast cancer or for chemoprevention up to 30 days following baseline visit (ok to initiate screening up to 2 months before planned baseline visit). Concurrent LHRH agonist, anti-HER2 directed therapy (e.g., trastuzumab, pertuzumab, ado-trastuzumab emtansine), and/or CDK4/6 inhibitor therapy (e.g., palbociclib, ribociclib, abemaciclib) is permitted. Prior tamoxifen and/or toremifene is permitted.
* Completion of surgery (mastectomy or lumpectomy/partial mastectomy) for treatment of breast cancer. Completion of axillary surgery as indicated (not required). For patients at high risk of breast cancer who have not been diagnosed with breast cancer, no surgery is required.
* Completion of chemotherapy, if indicated. Concurrent use of radiation therapy, LHRHa therapy, anti-HER2 therapy, PARP inhibitor, and CDK4/6 inhibitor therapy is permitted. Prior tamoxifen is permitted.
* Agree to avoid taking omega-3 fatty acid supplements from sources outside the trial during study participation.
* ECOG Performance Status ≤ 3.
* Able to complete questionnaires in English.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria

* Prior use of AI therapy for treatment or prevention of breast cancer.
* Use of omega-3 fatty acid supplementation during the 3 months prior to enrollment. Consumption of O3-FA through diet is permitted.
* Use of warfarin, enoxaparin, or direct oral anticoagulants within 7 days prior to registration.
* Known chronic liver disease (laboratory studies will not be assessed). Patients with hepatosteatosis, viral hepatitis, or other liver disorders who have adequate liver function according to the treating physician are permitted to enroll.
* Known symptomatic paroxysmal atrial fibrillation or persistent atrial fibrillation (EKGs will not be performed).
* History of pancreatitis.
* Hypersensitivity to fish and/or shellfish.
* Unable to take oral medications.
* Any medical condition that would interfere with the absorption of study medication capsules.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not, in the opinion of the treating investigator, have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Change in percentage of total fatty acids for each polyunsaturated fatty acid (PUFA) group from start of Omega-3 Fatty Acid (O3-FA) supplementation to 3 months of O3-FA | From start of Omega-3 Fatty Acid (O3-FA) supplementation to 3 months of O3-FA (at 6 months after start of AI therapy)
  Plasma oxylipins from blood samples collected at the start of O3-FA supplementation (3 months after start of Aromatase Inhibitor [AI] therapy alone) and after 3 months of AI therapy + O3-FA supplementation (6 months after start of AI therapy alone) will be quantified using solid phase extraction-liquid chromatography-electrospray ionization tandem mass spectroscopy. Oxylipins will be grouped according to PUFA substrate (linoleic acid [LA], arachidonic acid [AA], alpha-linoleic acid [ALA], eicosapentaenoid acid [EPA], and docosahexaenoic acid [DHA]). For each patient, the percentage of total fatty acids of each PUFA group will be calculated at both time points. The overall study percentage per PUFA group will be derived from the mean percentage of that PUFA group for all patients at each time point. The change in percentage between the two time points will be reported in tabular format for each PUFA group.

SECONDARY OUTCOMES:
Change in percentage of total fatty acids for each PUFA group from baseline to 6 months of Aromatase Inhibitor (AI) (3 months of AI alone + 3 months of AI with O3-FA supplementation) | At 6 months after start of AI therapy
  Plasma oxylipins from blood samples collected at baseline (before AI therapy) and at 3 months of AI therapy + O3-FA supplementation (O3-FA supplementation starts 3 months after start of AI therapy) will be quantified using solid phase extraction-liquid chromatography-electrospray ionization tandem mass spectroscopy. Oxylipins will be grouped according to PUFA substrate (LA, AA, ALA, EPA and DHA). For each patient, the percentage of total fatty acids of each PUFA group will be calculated at both time points. The overall study percentage per PUFA group will be derived from the mean percentage of that PUFA group for all patients at each time point. The change in percentage between the two time points will be reported in tabular format for each PUFA group.
Change in percentage of total fatty acids for each PUFA group from baseline to 3 months of AI therapy alone | At 3 months after start of AI therapy
  Plasma oxylipins from blood samples collected at baseline and at 3 months after start of AI therapy alone will be quantified using solid phase extraction-liquid chromatography-electrospray ionization tandem mass spectroscopy. Oxylipins will be grouped according to PUFA substrate (LA, AA, ALA, EPA and DHA). For each patient, the percentage of total fatty acids of each PUFA group will be calculated at both time points. The overall study percentage per PUFA group will be derived from the mean percentage of that PUFA group for all patients at each time point. The change in percentage between the two time points will be reported in tabular format for each PUFA group.
Number of participants who develop AI-associated musculoskeletal symptoms (AIMSS) | Up to 9 months after start of AI therapy
  Patients will be considered to have developed AIMSS if any of the following apply: (1) a ≥0.22 increase in the Health Assessment Questionnaire (HAQ) score within 9 months, (2) a ≥2.0 increase in Brief Pain Inventory (BPI) average pain within 9 months, or (3) discontinuation of AI therapy within 9 months because of new or worsened musculoskeletal symptoms, assessed using a protocol-specific discontinuation form completed by the patient's provider. The HAQ assesses interference of pain with daily activities (range 0-3), with change of 0.22 defined as a clinically meaningful difference, as noted in the literature.* The BPI assesses average pain over 7 days (range 0-10), with a change of 2.0 defined as a clinically meaningful difference, as noted in the literature.* Patients whose providers specify pain as the first or second-ranked reason for discontinuation will be considered to have discontinued AI therapy because of new or worsened musculoskeletal symptoms. *See references.
Number of participants that discontinue AI therapy due to AIMSS | Up to 9 months after start of AI therapy
  Patients whose providers specify pain as the first or second-ranked reason for discontinuation (in a protocol-specific discontinuation form) will be considered to have discontinued AI therapy because of new or worsened musculoskeletal symptoms.
Number of participants that discontinue AI therapy due to toxicity. | Up to 9 months after start of AI therapy
  Patients whose providers specify toxicity as the first or second-ranked reason for discontinuation (in a protocol-specific discontinuation form) will be considered to have discontinued AI therapy due to toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Henry, MD, PhD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolfe F, Michaud K, Strand V. Expanding the definition of clinical differences: from minimally clinically important differences to really important differences. Analyses in 8931 patients with rheumatoid arthritis. J Rheumatol. 2005 Apr;32(4):583-9. PMID 15801011
- [Background] Farrar JT, Pritchett YL, Robinson M, Prakash A, Chappell A. The clinical importance of changes in the 0 to 10 numeric rating scale for worst, least, and average pain intensity: analyses of data from clinical trials of duloxetine in pain disorders. J Pain. 2010 Feb;11(2):109-18. doi: 10.1016/j.jpain.2009.06.007. Epub 2009 Aug 8. PMID 19665938